CLINICAL TRIAL: NCT05234359
Title: Rapid Research in the CHILD Cohort to Inform Canada's Response to the COVID-19 Pandemic: Investigating the Prevalence & Predictors of SARS-CoV-2 Infection and the Health & Psychosocial Impact of the COVID-19 Pandemic on Canadian Families.
Brief Title: The CHILD Cohort COVID-19 Add-On Study
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Research Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: VR5 - 172658; 02207-000, 02205-000 (Other Grant/Funding Number: Research Manitoba (Winnipeg))
Record Dates: First submitted 2022-01-10; First posted 2022-02-10 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: COVID-19 pandemic; SARS-CoV-@ infection susceptibility and severity; pediatrics; mental health and wellbeing; seroprevalence; immunology; epidemiology; viral infection history; CHILD Cohort Study; data integration
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Psychological Well-Being | interventions — COVID-19 Serological Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — * Blood samples will be taken for SARS-Cov2 lgG serology testing.
  * Saliva samples collected for genetic and viral analysis and for antibodies, microbiota and hormones.
  * Stool samples collected for genetic, microbial and viral analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHILD Cohort Study: CHILD Cohort Study, a general population cohort of 3500 families (n~12,000) with children born in BC, AB, MB and ON between 2009-12. CHILD has dense longitudinal data (pregnancy to children aged 5-8 years) on physical and mental health, emotional wellbeing, child behaviour problems, and parenting stress, providing the powerful opportunity to identify and study changes in these parameters during the pandemic. CHILD participants have also granted permission for data linkage, providing the opportunity to link study data with administrative health data including clinical diagnoses, hospitalization and medication use. In this grant, the investigators will monitor SARS-CoV-2 seroprevalence among CHILD families and collect information about how they are experiencing the COVID-19 pandemic over the next 12 months.
  Interventions - Diagnostic Testing via home kit at 2 timepoints:
  Blood sample, Saliva sample, Stool sample
  Interventions: Diagnostic Test: Serology Testing; Diagnostic Test: Stool sample

INTERVENTIONS:
Diagnostic Test: Serology Testing — A simple home sampling kit containing volumetric absorption microsampling devices (Mitra(R) cartidge device, Neoteryx LLC) will be used by the participants to collect a finger stick blood sample (10 ul; a few drops). Kits will be delivered to participants' homes and returned by mail. An instructional video will be provided.
  Other Names: Blood samples; Finger stick blood sample
Diagnostic Test: Stool sample — Stool samples collected for genetic, microbial and viral analysis.

SUMMARY:
The objective of this study is to determine the prevalence and transmission of SARS-CoV-2 infection among Canadian children and parents in the CHILD cohort, identify predictors of infection susceptibility and severity, and understand the health and psychosocial impacts of the COVID-19 pandemic on CHILD families.

DETAILED DESCRIPTION:
Study will leverage the existing CHILD Cohort Study. All household members from each family will be incited to participate. To accommodate institutional physical distancing policies, the study is designed to minimize participant contact and the need for research staff onsite.

Weekly symptom check (by text message): Brief survey will capture COVID-19 signs and symptoms, testing and results, and healthcare utilization. Questions will be aligned with the Government of Canada self-assessment tool and harmonized with international partners.

Quarterly CoRonavIruS Health Impact Survey (CRISIS) (7) and body weight: 10-minute CRISIS survey captures COVID-19 exposure, life changes due to the COVID-19 crisis, daily behaviours, emotions and worries, media use and substance use. Each household member will complete the survey; parents will complete on behalf of younger children. Body weight (measured at home) will also be reported.

Repeated seroprevalence survey: Use of simple home sampling kit containing volumetric absorption micro-sampling devices (Mitra(R) cartridge device, Neoteryx LLC) to collect a fingerstick blood sample (10 ul; a few drops) for SARS-Cov2 IgG serology testing laboratory. Knowledge Users (Public Health authorities) and virology/serology experts will advise on the best available serology assay at the time of testing, and the investigators will consider testing in a public health lab if possible. Kits will be delivered and returned by mail, and an instructional video will be provided. Results will be returned to participants with appropriate explanation of their clinical relevance, and shared in real time with Knowledge Users to inform modeling efforts and pandemic management The timing and frequency of sero-surveys will be guided by our Knowledge Users depending on the progression of the pandemic.

Analysis of recently-collected pre-pandemic bio-samples: To determine the pre-pandemic immune profile of CHILD index children, the investigators will analyze a subset including all cases (asymptomatic and symptomatic) detected by serology and symptom surveys, plus a random subset of uninfected controls (estimated: 400 children in total). The investigators will assess:

1. a panel of innate and adaptive cytokines and chemokines using a commercial multiplex assay,
2. immune cell phenotypes using high dimensional flow cytometry
3. viral antibodies to establish prior/recent infections and cross-reactivity using targeted ELISA assays developed for antibodies to other human beta-coronaviruses

ELIGIBILITY:
Inclusion Criteria:

* All study participants enrolled in the original CHILD Cohort study are eligible for this add-on study
* Individuals living in the same household as study participants enrolled in the original CHILD Cohort Study are also eligible for this add-on study

Exclusion Criteria:

* CHILD Cohort Study participants who have been previously withdrawn from the study are not eligible for this add-on study
* CHILD Cohort Study participants who have not agreed to future contact by the study team are not eligible for this add-on study
* Participants (with the exception of children) who are not able to provide consent on their own behalf are not eligible for this add-on study
* Participants (with the exception of children) who are not able to read, write and understand English are not eligible for this add-on study
* Participants residing outside of Canada will not be participating in the sample collection component of this study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will seek the participation of the original families recruited into the CHILD Cohort Study (child and one or both of their parents or guardians) and any additional interested members from the same household (e.g siblings, grandparents etc). The CHILD Cohort Study is a general population cohort of 3500 families (~12,000 individuals) with children born in BC, Alberta, Manitoba and Ontario. Pregnant mothers were recruited into the study in 2009-2012.
  Exclusion criteria for initial recruitment to the CHILD study was mothers pregnant with more than one baby, had in-vitro fertilization (IVF) to become pregnant, baby had severe health problems at birth or was born prior to 35 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 5385 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Real-Time data on SARS-CoV-2 infection, severity, transmission and immune response | Biweekly, up to 70 weeks from Dec 2020 through Mar 2022
  Weekly Symptom check (by text message) Brief survey will capture COVID-19 signs and symptoms, testing and results, and healthcare utilization. Questions will be aligned with the Government of Canada self-assessment tool and harmonized with international partners
Identify biological and sociodemographic predictors of SARS-CoV-2 infection | Quarterly (once every 3 months - total duration 12 months), from Dec 2020 through Mar 2022. Baseline survey (Dec - May 2021); Follow-up 1 Survey (July - Aug 2021); Follow-up 2 Survey (Oct - Dec 2021); Follow-up 3 (Jan - Mar 2022)
  Quarterly CoRonavIruS Health Impact Survey (CRISIS) (7) and body weight: The 10-minute CRISIS survey captures COVID-19 exposure, life changes due to the COVID-19 crisis, daily behaviours, emotions and worries, media use and substance use. Each household member will complete the survey; parents will complete on behalf of younger children. Body weight (measured at home) will also be reported.
Understand the psychosocial, health and equity impacts of the COVID-19 pandemic and its management on CHILD families, and identify equity impacts | Quarterly (once every 3 months - total duration 12 months), from Dec 2020 through Mar 2022. Baseline survey (Dec - May 2021); Follow-up 1 Survey (July - Aug 2021); Follow-up 2 Survey (Oct - Dec 2021); Follow-up 3 (Jan - Mar 2022)
  Quarterly CoRonavIruS Health Impact Survey (CRISIS) (7) and body weight: The 10-minute CRISIS survey captures COVID-19 exposure, life changes due to the COVID-19 crisis, daily behaviours, emotions and worries, media use and substance use. Each household member will complete the survey; parents will complete on behalf of younger children. Body weight (measured at home) will also be reported.
Determine pre-pandemic immune profile of CHILD index children | 12 months
  Analysis of recently-collected pre-pandemic bio-samples: To determine the pre-pandemic immune profile of CHILD index children, we will analyze a subset including all cases (asymptomatic and symptomatic) detected by serology and symptom surveys, plus a random subset of uninfected controls (estimated: 400 children in total). The investigators will assess: a) a panel of innate and adaptive cytokines and chemokines using a commercial multiplex assay, b) immune cell phenotypes using high dimensional flow cytometry and c) viral antibodies to establish prior/recent infections and cross-reactivity using targeted ELISA assays developed for antibodies to other human beta-coronaviruses

SECONDARY OUTCOMES:
SARS-CoV-2 infection, severity, transmission and immunity. Prevalence and severity of infection | 12 months
  Prevalence and severity of infection will be estimated in real-time from weekly reports, and confirmed from serology testing. Severity will be classified as asymptomatic, mild or severe using WHO criteria. Transmission will be assessed using a multilevel modeling approach by province, house, and individual. Persistence of potential immunity will be determined from longitudinal serology testing for SARS-CoV-2 antibodies.
Identify biological, health and sociodemographic predictors of SARS-CoV-2 infection susceptibility and severity | 12 months
  In addition to the new data generated by this grant, the investigators will access existing data from the CHILD database, which contains over 50 million data points including multi-omics measurements from biological samples; indoor exposures including tobacco smoke; longitudinal clinical data on cardiometabolic and respiratory health, anthropometrics and body composition; mental health and psychosocial data; health behaviour data including sleep, physical activity, screen time and diet; and socioeconomic data including ethnicity. CHILD data is also integrated with www.CANUE.ca environmental data including weather, air quality and population density data. The investigators will use two approaches to analyze these data: hypothesis-driven and unbiased machine learning.
Understand the psychosocial, health and equity impacts of the COVID-19 pandemic | 12 months
  The investigators will identify individuals experiencing a decline in mental or physical health during the pandemic (not due to infection) and identify families and individuals experiencing food insecurity, financial difficulties, domestic violence and substance abuse. The investigators will report the prevalence of these outcomes to our knowledge users monthly. The investigators will use hypothesis-driven and unbiased approaches to identify factors that may predict risk for - or resilience against - these negative impacts of the pandemic. The investigators will also investigate socioeconomic inequities.
Sex-and-gender-based analysis | 12 months
  Sex differences in COVID-19 severity have been reported in adults (8) and gendered health behaviours are relevant to exposure and transmission. Mental health effects may also vary by sex and gender. It is not known if these differences exist in children, and how they might affect asymptomatic infection and transmission. The investigators will disaggregate all analyses by sex and/or gender in order to address these issues.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Azad, PhD, Principal Investigator — University of Manitoba; Padmaja Subbarao, MD, Study Director — University of Toronto
Locations (1):
- SickKids - The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study data will be entered into REDCap and OpenSpecimen. Questionnaires/forms will only collect de-identified information using the study number. When the questionnaires/ forms collect postal code, the fields will be flagged as containing identifying information. Names and email addresses will be used to send out online questionnaire reminders to participants. All other identifying information will be stored separately from study data, password protected and accessed only by local staff who contact participants. Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the NCC. This will not include the participant's contact or identifying information. Questionnaire and analyzed data, once cleaned will be de-identified and shared with other approved research team members. At the end of the study, all study databases will be de-identified and archived at the NCC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study data will be retained indefinitely.
Access Criteria: All IPD will be kept behind two security measures or as per equivalent institutional policy, under the supervision of the site Principal Investigator and will not be transferred outside of the study site. The study monitor, auditor and representatives of the Research Ethics Board (REB) may inspect all documents and records required to be maintained by the Principal Investigator, including but not limited to, medical records for the participants in this study. The study site will permit access to such records. Access to stored samples at the laboratory will be limited to the approved research team. When the study is completed, access to the de-identified, archived study data and/or samples will be provided through the CHILDdb (database).